CLINICAL TRIAL: NCT01197599
Title: Acute Tendon and Nerve Responses to Exercise
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Other Study IDs: TMP-MN-003
Record Dates: First submitted 2010-08-18; First posted 2010-09-09 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Cord Injury
Keywords: Healthy Control
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spinal Cord Injury
- Able-Bodied Control

SUMMARY:
The purpose of this study is to use ultrasound to analyze the effects of a bout of circuit training on the upper extremity of persons with spinal cord injury and able-bodied controls.

DETAILED DESCRIPTION:
Background: Manual wheelchair propulsion is a primary source of mobility for many individuals with spinal cord injury (SCI). Propelling a manual wheelchair over an extended period often leads to arm pain and, subsequently, to secondary disability. Over 50% of manual wheelchair users with SCI experience arm pain that limits their activities of daily living. The prevalence of shoulder pain and carpal tunnel syndrome among manual wheelchair users is between 31% and 73%, and 49% and 73% respectively. A circuit training protocol has been developed to strengthen and protect the muscles of people with SCI, and has been shown to improve muscle strength and endurance, and reduce HDLcholesterol levels.

Purpose: The purpose of this study is to use ultrasound to analyze the effects of a bout of circuit training on the upper extremity of persons with SCI and able-bodied controls.

Hypotheses: All subjects will show an increase in nerve cross-sectional area after participation in the circuit training protocol. Nerves and tendons will become less echogenic after participation in the circuit training protocol. These changes will be more pronounced in persons with SCI.

Methods: Data collected will include history of pain, a physical exam, and ultrasound images of the nondominant upper extremity before and after a bout of circuit training, which includes exercises lifting weights and using an arm cycle. Before circuit training, ultrasound images will be collected once. After the circuit training, ultrasound images will be collected every 10 minutes over an hour. These images and will be used to measure the health and properties (such as size) of nerves, muscles, and tendons in the arm. Changes in these properties after a bout of circuit training will be related to history and physical exam information.

ELIGIBILITY:
Inclusion Criteria:

Spinal Cord Injury Cohort:

* any cause or severity of spinal cord injury
* at least 1 year post-injury

Able-Bodied Control Cohort:

* self-reported good health

Exclusion Criteria:

* history of non-dominant traumatic upper extremity injury to both wrist and shoulder
* history of cardiopulmonary or other disease for which intense activity carries any risk of harm
* a progressive or degenerative disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample of persons with spinal cord injury or healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Nerve cross-sectional area | 1 day (Visit 1)
  Nerve cross-sectional area will be measured via ultrasound. Images will be collected at least once (pre-activity) and up to every 10 minutes over an hour (post-activity).

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami, The Miami Project to Cure Paralysis
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States